CLINICAL TRIAL: NCT04133012
Title: A Prospective Study Aiming to Determine the Cartography of Virological Reservoir Related to Antiretroviral Concentrations in Chronic HIV-1 Patients Treated with a First Line of Dolutegravir and Associated Nucleoside / Nucleotide Reverse Transcriptase Inhibitors (NRTIs).
Brief Title: Cartography of Virologic Reservoir Related to Antiretroviral Concentrations in HIV-1 Chronic Patients Treated by a First Line Treatment Containing Dolutegravir and Associated Nucleoside / Nucleotide Reverse Transcriptase Inhibitors Backbone
Acronym: DOLUVOIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ANRS EP64 DOLUVOIR
Record Dates: First submitted 2019-09-26; First posted 2019-10-21 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2023-08

CONDITIONS: HIV-1 Infection
Keywords: Viral cartography; Viral reservoir; Antiretroviral treatments diffusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Other): Single arm composed by 34 HIV-1 infected male subjects
  Interventions: Other: Samplings

INTERVENTIONS:
Other: Samplings — * blood samples
  * rectal biopsies
  * nodes biopsies
  * cutaneous fat tissues biopsies
  * semen sample

SUMMARY:
The main objective of the study is to characterize the diffusion of dolutegravir and associated backbone (abacavir/lamivudine or tenofovir/emtricitabine) in HIV-1 chronic patients in the main putative reservoirs, namely inguinal lymph nodes, rectal, fat tissues and sperm.

DETAILED DESCRIPTION:
The major obstacle to a functional cure of HIV infection is the persistence of the latent HIV reservoir.

Several arguments suggest the persistence of a residual viral replication in different compartments, despite an effective antiretroviral treatment. This residual viral replication partially comes from pharmacological sanctuaries where the drugs do not largely penetrate. In such sanctuaries a recent report published in Nature has shown that the virus can replicate with less antiviral pressure contributing to continuously replenish the reservoirs. Nevertheless, this study concerned a limited number of patients and only blood and lymph-node samples were collected for viral analysis. Moreover, the drug distribution was estimated based on mathematical hypotheses without drug measure concentration.

The International AIDS Society recommend for most patients an optimal initial regimen containing 2 nucleoside reverse transcriptase inhibitors (NRTIs) plus an integrase strand transfer inhibitor (InSTI)2. The new integrase inhibitor dolutegravir is more and more widely used in combination with nucleoside/nucleotide reverse transcriptase. Indeed, this drug shows a good tolerance and demonstrates a particularly fast inhibition of the viral replication. Moreover, dolutegravir is active against HIV strains that are resistant to the first generation of integrase inhibitors, raltegravir and elvitegravir. However the penetration of dolutegravir in deep compartments has not been fully characterized: the studies comprised a small number of patients and were not able to estimate the distribution in several compartments at the same time for each patient. Moreover the levels of residual viral replication in those compartments during treatment are unknown, making it difficult to evaluate the capacity of this drug and associated backbone to efficiently act against viral reservoirs maintenance.

The aim of the study is to measure simultaneously dolutegravir and nucleoside/nucleotide reverse transcriptase inhibitors in different compartments to obtain cartography of dolutegravir and associated backbone distribution and the spatial dynamics of virus in each patient.

The decision to study dolutegravir and the two associated backbones (abacavir / lamivudine or tenofovir /emtricitabine) was decided as:

* The International AIDS Society recommend for most patients an optimal initial regimen containing 2 nucleoside reverse transcriptase inhibitors (NRTIs) plus an integrase strand transfer inhibitor (InSTI)2.
* Dolutegravir viral power is established for high levels of viral load 90 and this drug is widely used.
* This study is very complementary of studies ANRS SIVART and ANRS 169 OPTIPRIM 2.
* Dolutegravir is combined with abacavir + lamivudine in a single-tablet and is largely prescribed.
* Raltegravir and elvitegravir will not be analysed because the number of recruited patients should be more important to obtain sufficient data and the feasibility would not be sure.

ELIGIBILITY:
Inclusion Criteria:

* Male HIV-1 infected subjects
* Age > or = 18 years old
* Currently receiving as first line therapy 7 days a week for at least 18 months with dolutegravir (at 50 mg once a day) and two nucleoside/nucleotide reverse transcriptase inhibitors (abacavir/lamivudine or ,tenofovir/emtricitabine) or

  * Receiving first-line therapy 7 days a week for at least 18 months with dolutegravir (50 mg once daily) + abacavir/lamivudine followed by dual therapy with dolutegravir + lamivudine for at least 6 months; or
  * Receiving first-line therapy 7 days a week for at least 18 months with dolutegravir + tenofovir / emtricitabine followed by dual therapy with dolutegravir + lamivudine for at least 6 months.
* HIV RNA currently <50 Cp/mL, , and <50 Cp/mL 6 months after treatment initiation and <50 Cp/mL confirmed at 12 months after treatment initiation
* Normal PT, APTT and platelet count values at screening
* Written and informed consent signed by the person and the investigator (no later than the day of pre-enrollment and prior to any examination carried out as part of the study (article L1122-1-1 of the Public Health Code)
* Person affiliated or beneficiary of a social security scheme (article L1121-11 of the Public Health Code) (State Medical Aid or AME is not a social security scheme)

Exclusion Criteria:

* Single HIV-2 infection
* Dolutegravir antiretroviral monotherapy
* Contraindication to biopsy, taking anticoagulant and antiplatelet drugs
* Hemophilia
* Symptomatic sexually transmitted infection
* Being under guardianship or trusteeship mandate for future protection
* Participation in another research involving the human person, of category 1 or 2,
* Associated treatments (Carbamazepine, Oxcarbazepine, Phenytoin, Phenobarbital, Rifampicin, St. John's Wort)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-06-09 (Actual)

PRIMARY OUTCOMES:
Characterization of the diffusion of dolutegravir and associated backbone (abacavir/lamivudine or tenofovir/emtricitabine) in sperm | At Day 0, At time T0 (before taking treatments)
  Dosage of the different antiretroviral drugs molecules in sperm
Characterization of the diffusion of dolutegravir and associated backbone (abacavir/lamivudine or tenofovir/emtricitabine) in lymph nodes | At Day 0, between T1 (maximum 3 hours after tacking treatments) and T3 (8 hours after taking treatments)
  Dosage of the different antiretroviral drugs molecules in lymph nodes
Characterization of the diffusion of dolutegravir and associated backbone (abacavir/lamivudine or tenofovir/emtricitabine) in fat tissues | At Day 0, between T1 (maximum 3 hours after tacking treatments) and T3 (8 hours after taking treatments)
  Dosage of the different antiretroviral drugs molecules in fat tissues
Characterization of the diffusion of dolutegravir and associated backbone (abacavir/lamivudine or tenofovir/emtricitabine) in rectal tissues | At Day 0, T1 (maximum 3 hours after taking treatment)
  Dosage of the different antiretroviral drugs molecules in rectal tissues

SECONDARY OUTCOMES:
Characterization of the level of the replication (RNA-HIV) and the level of infection (DNA-HIV) in the reservoirs | At Day 0
  Analyze and comparison of the level of viral transcription by measuring the cell-associated HIV- RNA in the different tissues and fluids: lymphoid, rectal, genital secretion, blood and fat biopsies as well as cerebrospinal fluid. Analyze and comparison of the reservoir level by measuring the cell-associated total HIV- DNA in the different tissues and fluids
Study of the spatial dynamics of viral quasi-species In the different reservoirs | At Day 0
  Analyze of the spatial dynamics of HIV-DNA and HIV-RNA from Lymphoid, rectal, genital secretion, blood, fat cells by phylogenetic analyses after sequencing Env HIV-DNA and HIV-RNA
Study of the mutations of resistance in the integrase gene | At Day 0
  Description of resistance mutations in Integrase gene which could be linked to suboptimal concentrations of dolutegravir
Description for each compartment of the relationship between exposure to therapeutic combinations and the level of infection / viral replication | At Day 0
  Characterization of the relationship between the concentration of dolutegravir and backbone drugs with the level of wild type viral replication in the different compartments. Analyze of the impact of backbone drugs associated to dolutegravir on viral level production. Correlation between the level of resistant virus replication and the exposure to dolutegravir and the backbone drugs. Evaluation by simulation the effect of different dosing regimen of dolutegravir (including higher doses) on the level of viral replication and on resistance

CONTACTS AND LOCATIONS:
Overall Officials: Antoine CHERET, Principal Investigator — CHU Pointe-à-Pitre/Abymes
Locations (8):
- France (8):
  - Antoine-Beclere Hospital, Clamart
  - Bicetre Hospital, Le Kremlin-Bicêtre
  - Saint Antoine Hospital, Paris
  - Bichat Hospital, Paris
  - Hotel Dieu Hospital, Paris
  - Necker Hospital, Paris
  - Pitie Salpetriere Hospital, Paris
  - Tourcoing Hospital, Tourcoing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.anrs.fr/fr